CLINICAL TRIAL: NCT05058937
Title: A Study to Examine the Clinical Value of Comprehensive Genomic Profiling Performed by Belgian NGS Laboratories: a Belgian Precision Study of the BSMO in Collaboration With the Cancer Centre - Belgian Approach for Local Laboratory Extensive Tumor Testing (BALLETT)
Brief Title: A Study to Examine the Clinical Value of Comprehensive Genomic Profiling Performed by Belgian NGS Laboratories: a Belgian Precision Study of the BSMO in Collaboration With the Cancer Centre
Acronym: BALLETT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Belgian Society of Medical Oncology (Other)
Collaborators: Illumina, Inc. (Industry); OncoDNA (Industry); PierianDx (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BSMO2020-2
Record Dates: First submitted 2021-09-06; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Solid Tumor; Metastatic Cancer
Keywords: Comprehensive genomic profiling; Next generation sequencing; Tumor mutational burden; Mircosatellite instability; Molecular tumor board; Targeted therapy; Immunotherapy; Actionable variants
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Comprehensive genomic profiling — TSO500 (523 genes + MTB + MSI)

SUMMARY:
The project, called "BALLETT" (Belgian Approach of Local Laboratory Extensive Tumor Testing), has a double goal: (1) show the relevance of broad molecular profiling to improve oncological patients care, (2) demonstrate that broad molecular testing can be performed in a decentralized setting by local diagnostics laboratories in a fully standardized and uniform way while complying with the highest quality standards.

This 2-year study involves the consortium of 9 cooperating Belgian NGS laboratories and will enroll 936 metastatic or locally advanced cancer patients coming from 13 different Belgian hospitals and cancer centers. Upon inclusion, all cancer patients will be offered 'comprehensive genomic profiling' (CGP) using Illumina's TSO500 NGS panel. This targeted NGS panel of 523 genes allows for the detection of single nucleotide variants, small indels, copy number variations and fusions, as well as for the determination of the 'tumor mutational burden' (TMB) and the 'microsatellite-instability' status (MSI). Both the wet lab execution of the CGP as well as the biological and clinical classification of the variants will be performed in a fully standardized way among the 9 participating Belgian local NGS laboratories.

The CGP results will be interpreted and discussed in the weekly meeting of the BALLETT national molecular tumor board (MTB), composed of oncologists, pathologists, molecular biologists, geneticists and bioinformaticians. The MTB will provide recommendations for targeted or immunotherapy based on the CGP results. Clinical Decision Support platforms OncoKDM (OncoDNA) and Clinical Genomics Workspace (PierianDx), both expert software that turns NGS data into actionable clinical information, will be used. The resulting therapy recommendation may consist of an approved therapy, a clinical trial, a medical need program or off-label use of cancer drugs. Treating physicians will receive the MTB recommendations and decide on the actual management of their patients. Reasons for not following the MTB recommendation will be registered.

The objectives of the project are:

1. To evaluate the clinical value of CGP in "real-world" practice in giving patients with advanced/metastatic solid tumours broader access to precision medicine
2. To describe the landscape of genomic alterations and quantify the actionable variants detected by comprehensive panel testing
3. To evaluate the number of actionable variants that would have been missed if the NGS analysis was limited to the reimbursed NGS panel (ComPerMed panel).
4. To assess the technical success of CGP
5. To standardize CGP data analysis, clinical interpretation, therapy recommendation and reporting among participating laboratories to the highest extent possible
6. To describe and to quantify the uptake of treatments and the inclusion in clinical trials recommended by the molecular tumour board guided by the CGP
7. To assess clinical benefit by calculating PFS ratio for individual patients (PFS on CGP-selected therapy/PFS on prior therapy) (null hypothesis: ≤ 15% of patient population has PFS ratio of ≥ 1.3)
8. To work in a multi-stakeholder approach to attract more innovative treatments and clinical trials in Belgium
9. To establish a Belgian genomic tumor database under the authority of the governmental 'Sciensano' thereby increasing public health knowledge in Belgium

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and above)
* Patients with metastatic solid tumours that are candidates for systemic therapy (early lines are preferred). Numbers will be capped for frequent tumour types (breast cancer: 120 patients, NSCLC: 120 patients, colorectal cancer: 120 patients). There will be a cohort of 150 patients with rare tumours or tumours with rare histology (Eur. J. Cancer 2011; 47: 2493-2511). Patients will be recruited as they appear in clinical practice.
* Life expectancy of > 12 weeks.
* Patient showing an Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2.
* Patients eligible for reimbursed NGS (cfr. indications NGS convention) will also be tested by the local NGS panel although this is not required if the CGP is ISO 15189 accredited. In that situation, the CGP is considered the local NGS. Patients that are not eligible for reimbursed NGS testing may only be tested by CGP.
* Patients must have enough tissue from a metastatic (preferred) or primary lesion biopsy for local testing and CGP testing, sufficient to extract a minimum of 80 ng DNA diluted in TE 1x and 40-80 ng (80 ng recommended) RNA diluted in RNA-grade water for TSO500 library prep. The nucleic acid extract must meet the quality requirements specified in the protocol (See "TruSight Oncology 500 (TSO500) workflow - Workflow instructions for participant laboratories"). The tissue should not be more than 2 years-old and fixed in 10% neutral buffered formalin. Availability of metastatic biopsies retrieved after a previous therapy line are mandatory for patients treated with therapies that are known to induce acquired mechanisms of resistance (EGFR TKIs in NSCLC, aromatase inhibitors in breast cancer, TKIs in GIST…). Bone biopsies that undergo decalcification are not allowed.
* Patients can only be enrolled if they are also concomitantly registered in the Precision-1 study and the investigator agrees to subsequent registration of CGP-driven treatment given and the investigator assessed outcome on this and prior treatment (PFS based on RECIST 1.1 evaluation).
* Patients able to provide written informed consent prior to enrolment into a potential subsequent clinical trial.

Exclusion Criteria:

* Life expectancy of less than 12 weeks.
* Inability to comply with protocol procedures.
* Known presence of severe hematopoietic, renal, and/or hepatic dysfunction (according to the local PI).
* No informed consent provided.
* Patient is not enrolled and followed as provided in Precision-1.
* Insufficient DNA/RNA quantity (<80 ng DNA, <40-80 ng RNA) and quality (dCq value >5 for DNA, DV200 value <20% for RNA), (See "TruSight Oncology 500 (TSO500) workflow - Workflow instructions for participant laboratories").

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 936 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number/prevalence of variants with clinical significance | through study completion, an average of 1 year
  Number/prevalence of variants with a classification of clinical significance Tier 1A or 1B (strong clinical significance) and Tier 2C and 2D (potential clinical significance) using CGP versus local NGS testing (if available) and/or versus minimally required ComPerMed panel.
  Tiering according to Li et al. AMP/ASCO/CAP. J Mol Diagn 19:4-23, 2017.
Number/prevalence of alterations by type (SNVs, CNVs, fusions) | through study completion, an average of 1 year
Description of patient journey | through study completion, an average of 1 year
  Percentage of patients with MTB recommendation categorized according to variant-therapy match scoring system, percentage of patients accessing genotype-informed treatment, turnaround time from CGP request to MTB recommendation, proportion of patients accessing molecular guided therapy or immune checkpoint inhibitors or combinations based on the result of CGP, timing of treatment initiation following MTB recommendation, proportion of deviations from treatment recommendations and reasons (rapid clinical deterioration, other protocol, patient ineligible, off-label treatment unavailable, clinical trial not feasible (e.g. physical distance), clinical trial not recruiting, physician's decision, patient's choice, …)

SECONDARY OUTCOMES:
Percentage of patients with successful CGP | through study completion, an average of 1 year
PFS ratio | through study completion, an average of 1 year
  PFS based on RECIST 1.1 evaluation of patients on the CGP recommended therapy and PFS ratio (PFS on CGP-selected therapy/PFS on prior therapy) (null hypothesis: ≤ 15% of patient population has PFS ratio of ≥ 1.3)
Number of participating NGS laboratories continuing CGP after the study | through study completion, an average of 1 year
  Including cost calculation and reimbursement data to support economic analysis (microcosting from the lab perspective and budget impact from the payer's perspective).

CONTACTS AND LOCATIONS:
Locations (12):
- Belgium (12):
  - ASZ Aalst, Aalst
  - ZNA, Antwerp
  - GZA, Antwerp
  - AZ Sint-Jan, Bruges
  - AZ VUB, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - Universitaire Ziekenhuis Antwerpen, Edegem
  - UZ Gent, Ghent
  - Jessa Ziekenhuis, Hasselt
  - UZ Leuven, Leuven
  - AZ Delta, Roeselare
  - AZ Turnhout, Turnhout

IPD SHARING:
Plan to Share IPD: No